CLINICAL TRIAL: NCT01610063
Title: A Pilot Study for the Evaluation of the Clinic-wide Impact of the Antidepressant Pharmacogenomic Algorithm in an Outpatient Clinical Setting
Brief Title: Evaluation of an Antidepressant Pharmacogenomic Algorithm in an Outpatient Clinical Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Assurex Health Home (Industry)
Responsible Party: Principal Investigator, Daniel K. Hall-Flavin, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-005610
Record Dates: First submitted 2012-05-25; First posted 2012-06-01 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Depression
Keywords: Algorithm; Depression; Assurex; GeneSight
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided (Experimental): A pharmacogenomic algorithm (GeneSight) guided treatment decisions for antidepressant medication selection and appropriate dosing.
  Interventions: Other: Pharmacogenomic algorithm
- Unguided (No Intervention): Treatment as usual

INTERVENTIONS:
Other: Pharmacogenomic algorithm — Genetic test results for 4 genes were put through algorithm and provided to physician for guidance prescribing medication.
  Other Names: GeneSight
  Arms: Guided

SUMMARY:
This was a study of a genotyping tool that reported on how subjects responded to medications and could be used in a community psychiatry practice to improve medication choice for depression. After the DNA test, an interpretive report was provided to the subjects' physicians. The hypothesis of this pilot study was that it was feasible to use this pharmacogenomic algorithm in a new setting to treat depressed subjects..

DETAILED DESCRIPTION:
Antidepressant medications are among the most widely prescribed medications. However, only 35% to 45% of depressed patients have a complete remission of their illness when initially treated with these medications. Consequently, the Mayo Clinic psychiatric pharmacogenomic team developed a pharmacogenomic algorithm designed to improve the effectiveness and safety of antidepressant medications by providing guidance in medication selection and appropriate dosing. This algorithm has been incorporated into a new genotyping interpretative report. The pharmacogenomic algorithm is based on genotyping both copies of four informative genes. These four genes are: 1) the Cytochrome (P450 2D6) gene; 2) the Cytochrome (P450 2C19) gene; 3) the Serotonin Transporter gene (SLC6A4); and 4) the Serotonin 2A receptor gene (5HTR2A). The trial took place at the Franciscan Skemp Healthcare System in La Crosse, Wisconsin over the course of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between the ages of 18 and 80.
2. Major depressive disorder or depressive disorder not otherwise specified as ascertained by a physician or mental health professional licensed to diagnose.
3. Patient is an outpatient and not in imminent need of inpatient hospitalization, or a discharging inpatient with scheduled follow-up with a Behavioral Health psychiatrist.
4. Patient has been referred to see a psychiatrist for optimum medication management.
5. Patient's Hamilton Depression Rating score is >14
6. Ability to read, understand and sign an informed consent document

Exclusion Criteria:

1. Serious medical illness (as ascertained via the initial triage screening process)
2. Patients with a diagnosis of Bipolar I disorder
3. Patients with a diagnosis of Schizophrenia or Schizoaffective disorder
4. Patients who are legally unable to consent to enrollment in the study (i.e. patients with legal guardians)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel K. Hall-Flavin, Principal Investigator — Mayo Clinic
Locations (1):
- Franciscan Skemp HealthCare, La Crosse, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at Franciscan Skemp Hospital in La Crosse, Wisconsin, a member of the Mayo Clinic Health System.
Pre-assignment Details: 233 male and female patients between the ages of 18 and 80 years with a primary DSM-IV diagnosis of major depressive disorder or depressive disorder not otherwise specified (NOS) were approached for consent. 3 patients refused consent. 3 participants failed to meet eligibility criteria.
Period: Overall Study
Arm/Group | Guided | Unguided
Started | 114 | 113
Baseline | 114 | 113
Completed 2-week | 97 | 105
Completed 4-week | 86 | 98
Completed 8-week | 72 | 93
Completed | 72 | 93
Not Completed | 42 | 20
Not completed — Lost to Follow-up | 42 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Guided | Unguided | Total
Number analyzed (Participants) | 114 | 113 | 227
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (12.8) | 44.0 (12.1) | 42.62 (12.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 77 | 146
  Male | 45 | 36 | 81
Region of Enrollment [Number; unit: participants]
  United States | 114 | 113 | 227

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Quick Inventory of Depressive Symptomatology (QIDS-C16) Score From Baseline
Description: The QIDS-C16 is a 16-item scale that is clinician-rated; it is designed to assess the severity of depressive symptoms. The QIDS-C16 total score ranges from 0-27. Scores ranging from 0 to 10 correspond with no to mild depression, while scores >/= 11 correspond to moderate to severe depression. A negative change indicates improvement in the subject's depression, and a positive change indicates a worsening of the subject's depression.
Time Frame: baseline, 8-week visit
Population: This analysis was performed on subjects who completed the study. There were 8 out of 72 patients in the guided arm and 12 out of 93 patients in the unguided arm who did not have assigned medication color in green/yellow/red. The number analyzed per row is indicated as (n=guided,unguided).
Measure: Mean (Standard Deviation); unit: Percentage change in depression rating
Arm/Group | Guided | Unguided
Number analyzed (Participants) | 72 | 93
Percentage change in depression rating
  Subjects in red category (n=16, 18) | -41.2 (31.7) | -11.0 (31.9)
  Subjects in green/yellow category (n=48, 63) | -48.4 (28.1) | -31.8 (29.8)
Statistical Analysis 1: Comparison: Guided vs Unguided; Comparison for QIDS-C16; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Percentage Change in Hamilton Depression Rating Scale (HAMD-17) Score From Baseline
Description: The HAMD-17 is a 17-item scale that evaluates depressed mood, vegetative and cognitive symptoms of depression, and co-morbid anxiety symptoms. The 17 items are rated on either a 5-point (0-4) or a 3-point (0-2) scale. In general, the 5 point scale items use a rating of 0=absent; 1=doubtful to mild; 2=mild to moderate; 3=moderate to severe; 4=very severe. The 3-point scale items use a rating of 0=absent; 1=probable or mild; 2=definite. The total HAMD-17 score ranges from 0 (not ill) to 52 (severely ill). A negative change indicates improvement in the subject's depression/anxiety symptoms, and a positive change indicates a worsening of the subject's depression/anxiety symptoms.
Time Frame: baseline, 8-week visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change in depression rating
Arm/Group | Guided | Unguided
Number analyzed (Participants) | 72 | 93
Percentage change in depression rating
  Subjects in red category (n=16, 18) | -42.2 (24.8) | -15.0 (20.9)
  Subjects in green or yellow category (n=48, 63) | -49.5 (28.4) | -35.6 (31.7)
Statistical Analysis 1: Comparison: Guided vs Unguided; Comparison between groups for HAMD-17; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

3. Secondary Outcome: Percentage Change in Patient Health Questionnaire-9 (PHQ-9) Score From Baseline
Description: The PHQ-9 is the nine item depression scale of the Patient Health Questionnaire. The PHQ-9 is based directly on the diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual Fourth Edition (DSM-IV). Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 (no symptoms) and 27 (severe symptoms) for depression. A negative change indicates improvement in the subject's depression symptoms, and a positive change indicates a worsening of the subject's depression symptoms.
Time Frame: baseline, 8-week visit
Population: There were 8 out of 72 patients in the guided arm and 12 out of 93 patients in the unguided arm who did not have assigned medication color in green/yellow/red. The number analyzed per row is indicated as (n=guided,unguided). One subject in the guided arm (green/yellow) did not complete the PHQ-9 questionnaire at 8 weeks.
Measure: Mean (Standard Deviation); unit: Percentage change in depression rating
Arm/Group | Guided | Unguided
Number analyzed (Participants) | 72 | 93
Percentage change in depression rating
  Subjects in red category (n=16, 18) | -46.3 (35.8) | -15.5 (31.4)
  Subjects in green/yellow category (n=47, 63) | -44.0 (39.9) | -20.7 (63.9)
Statistical Analysis 1: Comparison: Guided vs Unguided; Comparison for PHQ-9; Test type: Other; p = 0.002, t-test, 2 sided

4. Secondary Outcome: Percentage Change in Outcome by Bin Status and Treatment Group
Description: The Genesight algorithm presents recommendations for antidepressants and antipsychotics in "bin status" associated with colors. Green indicates "Use as Directed." Yellow indicates "Use with Caution." Red indicates "Use with Increased Caution and with More Frequent Monitoring." Definitions of the depression questionnaires are found in previous outcome measures. A negative change indicates improvement in the subject's depression/anxiety symptoms, and a positive change indicates a worsening of the subject's depression/anxiety symptoms.
Time Frame: baseline, 8-week visit
Population: All subjects were evaluated for a bin status, but not all the arms had subjects assigned to every bin status (green, yellow, or red). Bin status for each category title is reported as (n=Guided, Unguided).
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Guided | Unguided
Number analyzed (Participants) | 72 | 93
Percentage change
  %Change in HAMD-17 score, red (n=16, 18) | -42.2 (24.8) | -15.0 (20.9)
  %Change in HAMD-17 score, green/yellow (n=48,63) | -49.5 (28.4) | -35.6 (31.7)
  %Change in QIDS-C16 score, red (n=16,18) | -41.2 (31.7) | -11 (31.9)
  %Change in QIDS-C16 score green/yellow (n=48,63) | -48.4 (28.1) | -31.8 (29.8)
  %Change in PHQ-9 score, red (n=16,18) | -46.3 (35.8) | -15.5 (31.4)
  %Change in PHQ-9 score, green/yellow (n=47,63) | -44.0 (39.9) | -20.7 (63.9)

5. Secondary Outcome: Pharmacogenomic Report Utilization
Description: Physicians were directed to complete a survey for each participant detailing their experiences during the study period.
Time Frame: baseline, 8-week visit
Population: The medication changes of patients were recorded only for patients who completed the 8-week study (n=72,93 for guided and unguided arms). For each row below, the number of subjects analyzed is indicated by (n=guided, unguided) arms.
Measure: Number; unit: percentage of participants
Arm/Group | Guided | Unguided
Number analyzed (Participants) | 72 | 93
percentage of participants
  Overall med/dose changes (n=72, 93) | 76.8 | 44.1
  Med/dose changes in red bin subjects (n=16, 18) | 93.8 | 55.6

6. Secondary Outcome: Physicians' Perception of Participant's Satisfaction With Their Care
Description: Physicians reported on their perception of each participant's satisfaction with their care only for patients who completed the 8-week study. Physicians were directed to complete a survey for each participant detaining their experience during the study period.
Time Frame: 8-week visit
Population: Physicians completed surveys for 89 participants (96%) from the unguided group, and for 37 participants (51.4%) from the guided group. For each row below, the number of subjects analyzed is indicated by (n=guided, unguided) arms. For the first row, one of the physicians who completed the survey did not answer this question.
Measure: Number; unit: percentage of physicians
Arm/Group | Guided | Unguided
Number analyzed (Participants) | 37 | 89
percentage of physicians
  Very high patient satisfaction (n=37,88) | 40.5 | 14.8
  Physicians satisfied with care (n=37,89) | 94.6 | 61.8
  Very confident/confident med selection (n=37,89) | 91.9 | 61.8

7. Secondary Outcome: Responders at Week 8
Description: Definitions of the depression questionnaires are found in previous outcome measures. Definition of responder: a participant who had 50% or higher reduction in psychiatric score from baseline.
Time Frame: baseline, 8 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Guided | Unguided
Number analyzed (Participants) | 114 | 113
percentage of participants
  HAMD-17 | 43.1 | 26.9
  PHQ-9 | 50.7 | 31.2
  QIDS-C16 | 44.4 | 23.7

8. Secondary Outcome: Remitters at Week 8
Description: Definitions of the depression questionnaires are found in previous outcome measures. Definition of remitter: a participant with score less than or equal to certain value (HAMD-17 <=7, QIDS-C16<=5, PHQ-9<5).
Time Frame: baseline, 8 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Guided | Unguided
Number analyzed (Participants) | 114 | 113
percentage of participants
  HAMD-17 | 30.6 | 21.5
  PHQ-9 | 25.4 | 16.1
  QIDS-C16 | 26.4 | 12.9

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Guided | Unguided
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/113
Other Adverse Events (participants affected / at risk) | 0/114 | 0/113

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes